CLINICAL TRIAL: NCT03299465
Title: Yoga for Persistent Fatigue in the Survivors of Bone Marrow Transplantation: A Feasibility Study
Brief Title: Yoga for Fatigue in the Survivors of Bone Marrow Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mohamad Baydoun, PhD Candidate, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00130548
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Fatigue; Cancer
Keywords: bone marrow transplantation; yoga
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga arm (Experimental): A six-week restorative yoga intervention consisting of a weekly, 60-minute yoga group class led by a certified yoga instructor along with twice-weekly home practice using yoga DVD.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — This is a single arm study and all participants will be assigned to a six-week restorative yoga intervention. Restorative yoga sessions will consist of gentle physical poses (asanas), breathing control (pranayama), and relaxation (savasana).

SUMMARY:
Cancer-related fatigue (CRF) after hematopoietic cell transplantation (HCT) is a persistent problem that limits activities and causes distress. Considering the high prevalence of CRF among HCT survivors and the limitations of currently existing treatments, there is a pressing need for establishing safe and effective options for reducing CRF after HCT. Based on evidence supporting the use of yoga for CRF in non-HCT populations, yoga is one option worthy of evaluation for ameliorating CRF in HCT patients. Yoga is easy to implement, may be appealing to HCT patients, and can be self-administered, which would encourage long-term use and potentially lead to a better control of persistent CRF in HCT survivors. The primary aim of the proposed study is to assess the feasibility of a yoga intervention for HCT survivors with CRF. Outcomes from this feasibility study will provide the information needed to design a larger, adequately powered randomized controlled trial to evaluate yoga for CRF in HCT survivors. This study will employ a mixed-methods, single-arm, pretest-posttest design with focus groups. Twenty HCT survivors who report at least moderate fatigue will be recruited from the HCT clinic, Michigan Medicine. Participants will be enrolled in a six-week Restorative yoga program. The program will consist of a weekly, 60-minute yoga group class led by a certified yoga instructor along with twice-weekly home practice using yoga DVD.

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objective: To assess the feasibility of an organized yoga intervention for HCT survivors with CRF.

Hypothesis: A trial of yoga in the HCT survivor population will be deemed feasible if at least 75% of study subjects demonstrated protocol adherence rate of at least 80%.

Secondary Objectives:

- Explore participants' perceptions regarding yoga and physical activity

Hypothesis: HCT survivors will be positive about yoga and will express satisfaction with the yoga program, as will be shown during focus groups that will be held at the end of the yoga program.

- Evaluate the association between yoga practice and self-efficacy and self-regulation

Hypothesis: Adherence to yoga will be associated with higher self-efficacy and selfregulation scores.

- Evaluate the changes in CRF scores from baseline to the end of the yoga program.

Hypothesis: CRF scores at the end of the yoga program will be lower than CRF scores at baseline.

- Evaluate whether changes in CRF are associated with changes in depression, sleep disturbances, physical activity, and pain.

Hypothesis 5: Improvement in CRF will be associated with increased physical activity and decreased depression, sleep disturbances, and pain.

- Evaluate the safety of yoga practice in HCT survivors.

Hypothesis: Yoga will be considered as a safe intervention for CRF in HCT survivors as demonstrated by the absence of adverse events or serious adverse events related to or associated with yoga practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult HCT survivors as defined by being at least 100 days post autologous or allogeneic transplantation for a malignant disease. There is no restriction to enrollment by donor type, donor cell source, presence or absence of graft versus host disease.
* Age ≥ 18 years at the time of transplant.
* A history of persistent CRF as defined by a perception of general CRF for at least one month before enrollment.
* A history of at least moderate CRF as defined by a CRF score of 4 or more on a 10-point Visual Analog Scale.
* Participants who are deemed qualified for yoga movements according to the Yoga Qualifying Movements Screening Checklist (a checklist developed by researchers at the University of California, Los Angeles to promote yoga safety through assessing the eligibility of each patient)

Exclusion Criteria:

* A self-reported current practice of yoga or any other mind-body therapy, including but not limited to meditation or hypnosis therapy in the past 30 days prior to study enrollment.
* Subjects currently on supplemental oxygen support.
* Subjects currently receiving hemodialysis.
* Subjects currently admitted to an inpatient unit at Michigan Medicine.
* Subjects with an uncontrolled, active infection. Subjects with viremia (Cytomegalovirus or other) may be enrolled, provided they are on active therapy and at the discretion of the treating physician.
* Subjects who have relapsed after their autologous or allogeneic transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Practice log | Weekly during the six-week intervention period
  Yoga practice at home will be documented on a log sheet to be filled out by participants at the end of each practice week. We will check class attendance during the weekly telephone call with the study participants. We will use a log sheet to document in-class yoga practice and location of the yoga performance. At the end of the program, the number of yoga practice hours per participant will be tabulated. This number will be used to evaluate participants' adherence to yoga practice.

SECONDARY OUTCOMES:
Side-effects/adverse events log | Weekly during the six-week intervention period
  All subjects will be asked to complete a Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) weekly. The PRO-CTCAE questionnaire in this study includes a total of six items (numbness and tingling, dizziness, blurry vision, muscle pain, joint pain, others).
Multidimensional Fatigue Symptom Inventory | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The Multidimensional Fatigue Symptom Inventory-Short Form (MFSISF) will be used to measure fatigue in the past seven days. The MFSISF includes a total of 30 items that produce five subscales: general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor. All items have a possible score of 0 to 4, 0 representing "not at all" and 4 being "extremely".
PROMIS-SF-Fatigue | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The PROMIS-SF-Fatigue will be used to measure fatigue in the past seven days. The PROMIS-SF-fatigue is a unidimensional scale that measures general fatigue. It contains eight items with a possible score of 1 to 5 for each item.
Brief Pain Inventory - Short Form | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The Brief Pain Inventory - Short Form (BPISF) will be used to measure pain in the past 24 hours. The BPISF is a 9-item questionnaire used to evaluate the severity of a participants' pain and the impact of pain on the patient's daily functioning.
PROMIS-SF-depression | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The PROMIS-SF-depression will be used to measure depression in the past seven days. The PROMIS-SF-depression contains eight items with a possible score of 1 to 5 for each item (1: never, 5: always).
PROMIS-SF-sleep disturbance | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The PROMIS-SF-sleep disturbance will be used to measure sleep disturbance in the past seven days. The PROMIS-SF-sleep disturbance contains eight items with a possible score of 1 to 5 for each item.
Index of Self-Regulation Scale | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The Index of Self-Regulation Scale (ISR) is designed to measure individuals' level of self-regulation for health behaviors. The ISR contains nine items that produces three subscales: reconditioning, stimulus control, and behavioral monitoring.
Self-Efficacy for Managing Chronic Disease Scale | At baseline (before treatment) and within 10 days of the last in-class yoga session
  Self-efficacy will be measured using the Self-Efficacy for Managing Chronic Disease Scale (SEMCD). The SEMCD contains six items. Each item has a possible score of 1 to 10 (1: not at all confident, 10: totally confident).
PROMIS-SF- physical function | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The PROMIS-SF- physical function contains 12 items with a possible score of 1 to 5 for each item (1: unable to do, 5: without any difficulty). All items are reversely coded. The total score can range from 12 to 60 with higher scores indicating better physical function.
electronic pedometer | At baseline (before treatment) and within 10 days of the last in-class yoga session
  The electronic pedometer is an objective measure of physical activity. It is a simple, unobtrusive device that can be placed on the belt or waistband to count the number of steps taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No